CLINICAL TRIAL: NCT02242916
Title: In Silico Clinical Trial, Comparing State of the Art Photon Modalities With Proton and C-ion Therapy for Recurrent Head & Neck Tumors: A Multicentric Planning Study From the ROCOCO (Radiation Oncology COllaborative COmparison) Group
Brief Title: State of the Art Photon Therapy Versus Particle Therapy for Recurrent Head & Neck Tumors; a Planning Study
Acronym: ROCOCO
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: University of Pennsylvania (Other); Philipps University Marburg (Other); University Medical Center Nijmegen (Other)
Responsible Party: Sponsor
Other Study IDs: ROCOCO re-irradiation HN
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: reccurent Head and Neck tumors; re-irradiation; photon; proton; carbon-ion
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with recurrent HN tumors: Patients with recurrent Head and Neck tumors
  Interventions: Radiation: Photon therapy versus proton therapy; Radiation: Photon therapy versus C-ion therapy

INTERVENTIONS:
Radiation: Photon therapy versus proton therapy
Radiation: Photon therapy versus C-ion therapy

SUMMARY:
Given that the cost of proton therapy is considerably higher than that of conventional radiotherapy with photons, it is necessary to establish whether these higher costs are worthwhile in light of the expected advantages2,3,4. Thus, clear evidence of the situations in which proton therapy outperforms conventional photon treatment is needed. The investigators therefore aim to demonstrate through an in silico trial that proton therapy decrease the amount of irradiated normal tissue and, consequently, the risk of side effects in the surrounding normal tissue as well as the risk of secondary tumors. The same overall treatment time and an equal number of fractions will be used for both treatment modalities wherever possible. The most optimal technique for each individual patient, based on objective criteria related to limiting dose to normal tissue, will be prescribed by the institution concerned for each treatment option.

DETAILED DESCRIPTION:
The CTV to PTV margin will be determined by the individual institutes according to the treatment technique and treatment modality. For all treatment plans, modified ICRU 50 will be applied. The ICRU 50 recommendation is that 100% of the target volume (PTV) receives at least 95% of the prescribed dose. In this work, participants agree that D98 > = 95%, D2 < = 107%, cold (< 95%) and hot (> 107%) spots should be avoided in general, and that no hot spots will be allowed outside the PTV. The same overall treatment time (OTT) and an equal number of fractions will be used for all treatment modalities.

Treatment plans will be carried out using either photons, protons and C-ions for dose calculation for the indication H&N re-irradiation. A multicentric patient dataset, which can be found on a secured website5,6, will be used. The output databases with matrices including 3D delineation, the deliverable physical dose, RBE map, and BED/ EQD2 will be made available. To guarantee a similar set-up between the three treatments, similar dose distributions will be used. For C-ion treatment planning, a 20% uncertainty in the RBE values will be taken into account.

All treatment plans will be performed in centers that are already operating and have experience in treatment planning. Photon treatment plans will be carried out in Nijmegen en Maastricht, proton treatment plans at the University of Pennsylvania (UPENN) and the C-ion treatment plans at the University Hospital Marburg (UHM). For photons, all primary treatment plans were performed according to the planning procedure of each individual participating center by selecting the best available technique. The secondary photon treatment plan will be performed according predefined fractionation schedule and tumor dose. The proton treatment plans for H&N tumors will be planned with active beam delivery using IMPT and/or passive 4D beam delivery (PSPT). The C-ion treatment plans will be planned using a raster-scanning technique (IMIT).

All relevant OAR are delineated in the primary and secondary study set. GTV/CTV will be used accordingly to the actual treatment. New DVH's will be calculated for the added OAR. The secondary plan (i.e. re-irradiation plan) will be calculated again for the best currently available options for Photon, proton and C-ions. Between primary and secondary treatment there is a period of 1 to 5 years for all patients. To be on the save site a 30 % recovery of brainstem and spinal cord is assumed. There will not be a correction for fraction size. For practical reasons the location of the Dmax in the brainstem or spinal cord will not be taken into account. A maximal cumulative dose of 120 Gy will be accepted in the mandibular.

If the mandibular is part of the CTV in the first as well as in the second treatment, a higher dose will be accepted. A cumulative dose of max 120 Gy will also be accepted for the larynx , for the arytenoid is this 100Gy, unless the larynx is within the CTV for the first and second treatment than a higher dose will be accepted.

This means that for a total study population of 25 patients per tumor site and group at least 100 treatment plans will be carried out. All dose maps will be saved on the secure website as part of the database mentioned above.

Photon, proton and C-ion treatments will be compared based on dosimetric parameters on normal tissues such as mean parotic dose, etc. In addition, the NTCP for a fixed tumor dose or the same expected TCP will be determined. Cobalt Gy equivalent doses will be used when reporting the proton and C-ion dose. In the case of protons, a constant RBE value of 1.1 will be used for both the tumor and the normal tissues. The RBE of C-ions will be calculated based on the models used by the participating centers. The GSI in-house treatment planning system uses RBE values calculated on the basis of the local effect model (LEM). The LEM I (alpha/beta=2) is based on the radial dose distribution of each charged particle crossing into a cell nucleus, as well as on the radiosensitivity and repair capacity of the tissue. The TPSs used by UHM is also based on the LEM model. The model used at NIRS utilizes fixed RBE values that are dependent on the depth in the body, but independent of dose level or tumor type.

ELIGIBILITY:
Inclusion Criteria:

* Primary treatment:

  1. ≥ 50 Gy with curative intent (with or without chemo)
  2. CTV includes primary tumor and at least level II-IV
  3. Severe dental scatter artifacts or metal implants of unknown density will be excluded
  4. IMRT plan available
* Secondary treatment after ≥ 1 year, dose 70 Gy

  a. Severe dental scatter artifacts or metal implants of unknown density will be excluded
* Overlap of at least one OAR in primary and secondary treatment

Exclusion Criteria:

* Patients referred for postoperative radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with recurrent head and neck tumors
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Radiation exposure for organs at risk in H&N cancer patients | 7 weeks
  Radiation exposure for organs at risk in H&N patients treated with radiotherapy for recurrent tumors after primary radiotherapy. Results are based on in silico planning study which compares photon, proton and Carbon-ion treatments. The same biological radiation dose, fractionation schedule and tumor dose inhomogeneity is used. A wide range of OAR is included in this study, to be able to document doses to organs that are further away from the target volume, and also to quantify low doses to organs.

SECONDARY OUTCOMES:
Normal tissue complication probability (NTCP) for a fixed tumor dose | 3 years
  Based on the OAR radiation exposure, the Normal tissue complication probability (NTCP) for a fixed tumor dose or the same expected Tumor Control Probability (TCP) will be determined using dose response curves.

OTHER OUTCOMES:
Risk of secondary cancer | 10 years
  Risk of secondary cancer

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Eekers, Dr., Principal Investigator — Maastro Clinic, Dr Tanslaan 12, Maastricht, The Netherlands; Philippe lambin, prof, Dr, Study Director — Maastro Clinic, Dr Tanslaan 12, Maastricht, The Netherlands
Locations (1):
- Maastro Clinic, Maastricht, Netherlands